CLINICAL TRIAL: NCT01562873
Title: Phase II Study of Ruxolitinib (INCB018424) in Patients With PSTAT3+ Breast Cancer
Brief Title: Ruxolitinib in Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough responses to continue treatment.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nancy Lin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-024
Record Dates: First submitted 2012-03-20; First posted 2012-03-26 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: pSTAT3+
MeSH Terms: conditions — Breast Neoplasms | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ruxolitinib-Cohort A (Experimental): Patients received Ruxolitinib 25 mg twice daily for up to 12 cycles (cycle duration=28 days) until evidence of disease progression or unacceptable toxicity. Patients enrolled sequentially into two possible cohorts based on pStat3+ expression score by central testing: Cohort A - moderate to high positive status defined as a score of >/=5 by central testing or Cohort B - low positive status defined as a score of 3-4. Each cohort was evaluated with a 2 stage design. Cohort B only opened if 2 objective responses were observed in 1st stage Cohort A patients (n=21).
  Interventions: Drug: Ruxolitinib
- Ruxolitinib-Cohort B (Experimental): Patients received Ruxolitinib 25 mg twice daily for up to 12 cycles (cycle duration=28 days) until evidence of disease progression or unacceptable toxicity. Patients enrolled sequentially into two possible cohorts based on pStat3+ expression score by central testing: Cohort A - moderate to high positive status defined as a score of >/=5 by central testing or Cohort B - low positive status defined as a score of 3-4. Each cohort was evaluated with a 2 stage design. Cohort B only opened if 2 objective responses were observed in 1st stage Cohort A patients (n=21).
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib
  Other Names: INCB018424; Jakafi

SUMMARY:
Ruxolitinib is a drug which blocks the Janus tyrosine Kinase (JAK) signaling pathway. It is thought that this pathway might be important in certain types of breast cancer, and that blocking this pathway might lead to anti-cancer effects. This study is testing the effects of ruxolitinib in patients with breast cancer.

DETAILED DESCRIPTION:
Objectives:

Primary

* The primary objective of this two-stage, phase II study is to estimate the objective response rate to ruxolitinib in patients with metastatic or unresectable locally advanced breast cancer which is pStat3+ and which has progressed on at least one line of chemotherapy for advanced disease, and/or has recurred within 12 months of completion of neoadjuvant/adjuvant chemotherapy.

Secondary

* To describe the toxicity profile
* To evaluate clinical benefit rate (CR + PR + SD >/= 24 weeks)
* To estimate progression-free and overall survival

Exploratory

* To explore whether baseline hs-CRP level higher than the group median is associated with objective response
* To explore whether baseline IL-6 level higher than the group median is associated with objective response
* To describe hs-CRP level over time, and to describe the proportion of patients with a) hs-CRP > 3mg/L at baseline, on treatment, and at time of progression, and b) hs-CRP > 1mg/L at baseline, on treatment, and at time of progression
* To describe IL-6 level over time, and to describe the proportion of patients with IL-6 level above the upper limit of normal at baseline, on treatment, and at time of progression
* To describe pStat3 status by IHC in baseline metastatic biopsies
* To describe pStat3 status by IHC in on-study biopsies
* To describe pStat3 status by IHC in the time of progression biopsy samples
* To characterize archival and metastatic biopsy samples using triple immunofluorescence for CD44, CD24, and pStat3
* To characterize archival and metastatic biopsy samples using a previously characterized pStat3 gene signature
* To characterize circulating tumor cells (CTCs) for CD44, CD24, and pStat3 at baseline and time of progression

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer
* Must have known ER, PR and HER2 status
* Either, Triple Negative Metastatic Breast Cancer or
* Inflammatory Breast Cancer with any ER, PR HER2 status
* Availability of archival tissue specimen suitable for pStat3 testing
* Life expectancy of greater than 3 months
* Measurable disease by RECIST
* At least one prior chemotherapy regimen for treatment of metastatic breast cancer and/or recurrence within 12 months of completion of neoadjuvant/adjuvant chemotherapy or
* For patients with inflammatory breast cancer but no distant metastases, progression through standard neoadjuvant chemotherapy is required

Exclusion Criteria:

* Pregnant or breastfeeding
* Active brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib
* Clinically significant malabsorption syndrome
* Concurrent use of medications/substances that are strong inhibitors of CY3A4
* No uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from October 2012 through June 2014.
Pre-assignment Details: Patients must have had sufficient archival specimen for central pStat3 testing to be eligible.
Period: Overall Study
Arm/Group | Ruxolitinib-Cohort A | Ruxolitinib-Cohort B
Started | 21 | 0 (The observed number of objective responses in Cohort A was not sufficient for Cohort B to open.)
Completed | 0 | 0
Not Completed | 21 | 0
Not completed — Disease Progression per RECIST | 10 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Clinical Disease Progression | 9 | 0
Not completed — Clinical PD and adverse event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Arm/Group | Ruxolitinib-Cohort A
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 51 [36 to 72]
Gender [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
pStat3 Positive Status [Number; unit: participants]
  moderate to high positive | 21
  low positive | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate (ORR) was defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; Treatment continued until disease progression or unacceptable toxicity up to 12 cycles. Treatment duration was a median of 2 cycles range (1-5).
Population: The analysis dataset is comprised all enrolled patients.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | Ruxolitinib-Cohort A
Number analyzed (Participants) | 21
proportion of patients | 0.0 [0.0 to .133]

2. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) was defined as achieving complete response (CR), partial response (PR), or stable disease (SD) for 24 weeks or longer based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria. SD needed to be a minimum 24 weeks in duration.
Time Frame: as for outcome 1
Population: The analysis dataset is comprised all enrolled patients.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | Ruxolitinib-Cohort A
Number analyzed (Participants) | 21
proportion of patients | 0.0 [0.00 to 0.133]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death or date last known alive and estimated using Kaplan-Meier (KM) methods.
Time Frame: In long-term follow-up, patients were followed for survival every 4 months for up to 2 years. Median follow-up in this study cohort was 4.5 months (range 0.6-21.9).
Population: The analysis dataset is comprised all enrolled patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ruxolitinib-Cohort A
Number analyzed (Participants) | 21
months | 4.5 [2.9 to 10.2]

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or equivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically every 8 weeks on treatment through 12 cycles and in long-term follow-up every 4 months for up to 2 years. Median follow-up in this study cohort was 4.5 months (range 0.6-21.9).
Population: The analysis dataset is comprised all enrolled patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ruxolitinib-Cohort A
Number analyzed (Participants) | 21
months | 1.2 [0.97 to 1.84]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout the 12 cycles of treatment and at time of off-treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. Other AEs were defined as events with treatment attribution of possible, probable or definite and grades 1 or 2 per CTCAEv4.
Arm/Group | Ruxolitinib-Cohort A
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib-Cohort A (N=21)
Anemia (Blood and lymphatic system disorders) | 2
Aspartate aminotransferase increased (Investigations) | 2
GGT increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ruxolitinib-Cohort A (N=21)
BL101 (Blood and lymphatic system disorders) | 1/5
GI108 (Gastrointestinal disorders) | 1/5
GI123 (Gastrointestinal disorders) | 1/5
GI179 (Gastrointestinal disorders) | 1/5
GI216 (Gastrointestinal disorders) | 2/5
CN101 (General disorders) | 1/5
CN105 (General disorders) | 1/5
CN108 (General disorders) | 3/5
CN109 (General disorders) | 1/5
IN999 (Infections and infestations) | 1/5
IV129 (Investigations) | 1/5
IV137 (Investigations) | 1/5
MU112 (Musculoskeletal and connective tissue disorders) | 1/5
MU999 (Musculoskeletal and connective tissue disorders) | 1/5
NE145 (Nervous system disorders) | 1/5
PU113 (Respiratory, thoracic and mediastinal disorders) | 1/5
PU114 (Respiratory, thoracic and mediastinal disorders) | 1/5
DE999 (Skin and subcutaneous tissue disorders) | 1/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No